CLINICAL TRIAL: NCT06433401
Title: The Effect of Structured Transition Care Model Applied to Adolescents With Congenital Heart Disease on Transition Readiness, Self-Management Skills and Care Satisfaction
Brief Title: The Effect of Structured Transition Care Model Applied to Adolescents With Congenital Heart Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, tutkukırçı, Principal Investigator, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AnkaraYBU-SBF-TKT-01
Record Dates: First submitted 2024-05-23; First posted 2024-05-29 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Congenital Heart Disease in Adolescence
Keywords: Congenital heart disease; Adolescent; Transition care; Nurses
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: The study included two groups, an intervention group and a control group. Intervention group receiving transitional care training and control group receiving routine care.
Who Masked: Participant
Masking Description: Participants will not know which group they are in. They will be assigned to groups by simple simple random randomization method. Since the researcher was the one who provided the training, researcher blinding could not be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transition care group (Experimental): The transitional care group is a group that will receive a transitional care training consisting of a total of 3 modules in which the content is arranged for individualized needs with expert opinion from 10 faculty members working in the field of Child Health and Diseases Nursing.The education sessions will be conducted every months in sessions of approximately 35-40 minutes face-to-face in the training room allocated to the individual researcher.
  Interventions: Behavioral: Transitional care training with brochures, posters and slide training materials
- Control group (No Intervention): The control group is the group receiving routine care that continues the normal follow-up of the clinic without any intervention. However, in terms of compliance with ethical principles, the same training will be given to them upon their request after the research is completely completed.

INTERVENTIONS:
Behavioral: Transitional care training with brochures, posters and slide training materials — Education at 1 and 2 months after the first interview
  Arms: Transition care group

SUMMARY:
Congenital heart disease is one of the most common congenital defects with a high mortality and morbidity rate. Children with congenital heart disease step from pediatric care to adult care during adolescence. This situation has brought up transitional care, which is defined as "the purposeful and planned movement of adolescents and young adults with chronic physical and medical conditions from pediatric to adult-oriented health systems". Since adolescents with congenital heart disease are at high risk for complications in adulthood, it is very important to raise awareness, increase the level of readiness for adult care and gain self-management skills during the transition phase. This study was planned as a randomized controlled experimental study to evaluate the effect of the developmental transition care model applied to adolescents with congenital heart disease during the transition from pediatric care to adult care on the transition readiness level, self-management skills and care satisfaction of adolescents.

Studies have shown that both adolescents with congenital heart disease and their caregivers need professional support, appropriate transition education and care before transition to adult care in order to increase adaptation to adult care, to gain self-management skills and to reduce their concerns. Studies in which adolescents are followed up after transition to adult care show that when the transition process is not successfully completed, there is excessive time between the last pediatric control and the first adult control or there are losses in further follow-up. Although there are studies in our country in which transition care is applied, this study is planned because there is no intervention study in which developmental transition care model is applied to adolescents with congenital heart disease. It is thought that this study will increase the transition readiness levels, self-management skills and care satisfaction of adolescents with congenital heart disease and guide the nurses working with them.

DETAILED DESCRIPTION:
Congenital heart disease is one of the most common congenital defects with high mortality and morbidity rates. The American Heart Association reports that at least eight out of every 1000 babies born are born with heart disease. In Turkey, an average of 11,000-17,000 babies are born with congenital heart disease each year. Congenital heart diseases are a very large group of diseases and the level and prognosis of defects in this group vary. While severe defects result in neonatal and infant mortality, almost all children with mild defects survive. With the adolescent period, children step from pediatric care to adult care. While the transition to adulthood causes psychological and social changes for a healthy adolescent and his/her family, the need for additional care for adolescents with chronic diseases and the change in access to health services make the transition period even more challenging. This situation has brought transition care, defined as "the purposeful and planned movement of adolescents and young adults with chronic physical and medical conditions from pediatric health systems to adult-oriented health systems" to the agenda. Since adolescents with congenital heart disease are at high risk for complications in adulthood, raising awareness of the need for regular medical follow-up and preparing them for changes in the health care environment are very important for a successful transition.

The aim of transitional care is to maintain the control and well-being of the disease in adulthood and maximize its potential by providing the quality care practices needed by the adolescent without interruption. Studies have shown that both adolescents with congenital heart disease and their caregivers need professional support, appropriate transition education and care before transition to adult care in order to increase their adaptation to adult care, gain self-management skills and reduce their concerns. The American Academy of Pediatrics (APA) recommends that the transition process should begin with transition planning between the ages of 12-14. However, since physiological and psychological development and needs are not related to the chronological age of the individual, the essence of timing in the transition process is flexibility. The timing of transition varies depending on many individual and environmental variables such as age, gender, physical and psychological maturation, current medical condition, compliance and adherence to treatment, readiness of the adolescent for transition, finding an appropriate adult care provider, and insurance policies. In studies in which adolescents with congenital heart disease were followed up after transition to adult care, when the transition process was not successfully completed, there was a gap between the last pediatric control and the first adult control. In conclusion, there is no intervention study in our country in which the developmental transition care model was applied to adolescents with congenital heart disease and the results were evaluated. In addition, based on clinical experiences and observations, it was determined that adolescents and their parents had difficulties in the transition from pediatric care to adult care and this negatively affected self-management related to the disease. The aim of this study was to evaluate the effect of the developmental transition care model applied to adolescents with congenital heart disease during the transition from pediatric care to adult care on the transition readiness level, self-management skills and care satisfaction of adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agree to participate in the research
* To be between the ages of 16-20,
* Having a diagnosis of congenital heart disease,
* Being followed up with a diagnosis of congenital heart disease for at least one year in the polyclinics where the study was conducted,
* To be able to communicate in Turkish,
* Not having any mental deficiency that may prevent communication

Exclusion Criteria:

* Refusing to participate in the research,
* Not being able to communicate in Turkish,
* Not showing up regularly for follow-ups,
* Having any mental disability that may prevent communication

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Transition Readiness Assessment Scale | at certain intervals for 1 year
  It addresses the readiness of adolescents/young adults with chronic diseases to transition from pediatric care to adult care with the sub-dimensions of management of treatment, management of appointments, monitoring of health status, communication with health personnel and management of daily activities. The Cronbach alpha internal consistency coefficient of the Turkish scale was .88. The readiness for transition assessment scale is a 5-point Likert-type self-assessment scale to assess the skills and behaviors required for disease management in five sub-dimensions. Each item is evaluated between 1 point (no, I do not know how to do it) and 5 points (yes, I can do it when I need to). Adolescents score a minimum of 20 and a maximum of 100 points. The higher the score obtained from the scale, the higher the level of readiness of the adolescent to transition from pediatric care to adult care.

SECONDARY OUTCOMES:
Data Collection Form on Sociodemographic and Medical Characteristics | at certain intervals for 1 year
  This form was prepared by the researchers as a result of the literature review and will be used to obtain information on the age, gender, contact information, information on parents interested in health checks, initial diagnosis characteristics (date of diagnosis and complaints of hospital admission), degree of congenital heart disease, information on regularly used medication, body mass index, physical activity status, nutritional status, vital signs, cardiac examination and imaging information of adolescents.
Chronic Disease Self-Management Scale | at certain intervals for 1 year
  This scale to determine the disease management skills of individuals with chronic diseases The scale consists of 21 items and 4 sub-dimensions. These sub-dimensions are self-stigmatization, coping with stigmatization, health care effectiveness and treatment compliance. It was stated that the scale is suitable for use in all individuals with chronic diseases. The scale score is calculated by arithmetic mean. Each item in the scale is scored between 1 and 5. Scores obtained from the scale indicate that self-management increases as it approaches 5, and self-management decreases as it decreases towards 1.
Transitional Care Satisfaction Rating Scale | at certain intervals for 1 year
  The scale allows adolescents with chronic diseases to self-assess the care they receive and to determine their expectations; it is a scale that addresses the care provided with the dimensions of "Management of the Physical Environment (PME)", "Health Personnel Characteristics (HCP)" and "Care Process (CP)". The form of the scale used for adolescents consists of two separate questionnaires (ideal care/existing care) with 21 questions in which the adolescent's expected care and current care are evaluated. The scale forms are 7-point Likert-type with 1=strongly disagree and 7=strongly agree. Participants are asked to rate their current care based on the best care they expect for themselves. Scoring is based on the difference between the individual's expectations and what they actually perceive.

CONTACTS AND LOCATIONS:
Overall Officials: Tutku KIRÇI TEMİZ, PhD s., Principal Investigator — Ankara Yildirim Beyazıt University; Evrim KIZILER, Asst.Prof., Study Director — Ankara Yildirim Beyazıt University; Utku ARMAN ÖRÜN, Prof.Dr., Study Director — Republic of Turkey Ministry of Health Ankara Etlik City Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Republic of Turkey Ministry of Health Ankara Etlik City Hospital, Ankara, Ankara Yenimahalle
  - Republic of Turkey Ministry of Health Ankara Etlik City Hospital, Ankara

IPD SHARING:
Plan to Share IPD: No